## ClinicalTrials.gov ID: NCT03659032

Efficacy of Pediatric Manual Therapy in the Positional Plagiocephaly

**Consent Form** 

Date: 09/01/2018

## **CONSENT FORM**

Doctoral Program in Health and Sport Sciences University of Zaragoza

| To be filled out by the examiner | |
|---|---|
| ID Number | |
| representative of the patient), acting as relationship with the patient: father, mother(name of the patient) | , etc.) of |
| I have read the information sheet that has been given to me. I have had the opportunity to ask any questions about the treatment. Any questions that I have asked have been answered to my satisfaction. I have received enough information about the treatment. | |
| I have talked to (name of the physical therapist in charge). | |
| I understand that the patient that I represer | erstand that the patient that I represent agrees to the treatment strategy. |
| I understand that the patient that I represent may withdraw from the study: 1 at any time | |
| 2 without explanation 3 without consequence or the treatment of the patient that I represent | - |
| I consent voluntarily for (name of the patient) to receive the treatment strategy developed in the plagiocephaly study. | |
| Signature of legal | |
| representative of the patient | Signature of researcher |
| Name: Date: | Name: Date: |